CLINICAL TRIAL: NCT02168699
Title: Ultrasound Imaging of Musculocutaneous Nerve in Infants, Preschoolers and Children
Brief Title: Ultrasonographic Detection of Musculocutaneous Nerve in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Paraskevi Matsota, MD, PhD, Attikon Hospital
Other Study IDs: ATTIK12112
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Sonographic Detection of Musculocutaneous Nerve
Keywords: children; infants; musculocutaneous nerve; ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultrasound examination (Other): Ultrasound examination of the axillary region in children
  Interventions: Other: Ultrasound examination of the axilla

INTERVENTIONS:
Other: Ultrasound examination of the axilla

SUMMARY:
Localizing the musculocutaneous nerve for neural blockade is crucial to achieve complete anesthesia of the forearm. However, in pediatric anesthesiology, the musculocutaneous nerve is unable to be blocked in up to 40-50% of cases when only neurostimulation is used, while there is limited information regarding ultrasound imaging of the musculocutaneous nerve in children.

The aim of this prospective imaging study is to investigate whether musculocutaneous nerve is visualized in childhood with the use of ultrasound imaging or not. A secondary aim of this study is to assess the percentage of its visualization according to the age.

Parental written informed consent is obtained from all participants. The children are divided into three groups according to their age: Group 1, with infants aged less than 12 months; Group 2, with toddlers and preschoolers; and Group 3, with school-aged children (6.5-12 years).

Children are placed in the supine position with the involved arm abducted at 90° and the elbow flexed at 90°. The linear probe of a portable ultrasound machine is placed at the axillary region, perpendicularly to the axillary artery. The musculocutaneous nerve is searched near the axillary artery (proximally) and its course is followed distally (into the coracobrachialis muscle). Its sonographic detection is recorded in these two sites, both proximally and distally.

ELIGIBILITY:
Inclusion Criteria:

* children 0-12 years old
* parental written informed consent

Exclusion Criteria:

* parental refusal
* children refusal
* previous operations to the axilla
* anatomical malformations of the axilla
* spasticity
* morbid obesity.

Max Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 2010-12; Primary Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Assession of the ultrasonographic visualization rate of musculocutaneous nerve in children | Data is assessed during sonographic examination of the axillary region

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of Anesthesiology, Attikon University Hospital, Athens, Attica, Greece